CLINICAL TRIAL: NCT00357461
Title: A Randomized Phase II Study of Fixed Dose Ipilimumab (MDX-010) 10 mg/kg Given Alone or in Combination With Two gp100 Peptides Emulsified With Montanide ISA-51 VG for Previously Treated HLA-A * 0201 Positive Subjects With Stage IV Melanoma
Brief Title: Ipilimumab With or Without Vaccine Therapy in Treating Patients With Previously Treated Stage IV Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000486705; NCI-06-C-0159; NCI-P6951; MDX-NCI-06-C-0159; NCT00325052 (obsolete NCT alias)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Protein Subunit Vaccines; incomplete Freund's adjuvant; Ipilimumab

INTERVENTIONS:
Biological: gp100:209-217(210M) peptide vaccine
Biological: gp100:280-288(288V) peptide vaccine
Biological: incomplete Freund's adjuvant
Biological: ipilimumab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as ipilimumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Vaccines made from gp100 peptides may help the body build an effective immune response to kill tumor cells. Giving ipilimumab together with vaccine therapy may be an effective treatment for melanoma.

PURPOSE: This randomized phase II trial is studying ipilimumab and vaccine therapy to see how well they work compared to ipilimumab alone in treating patients with previously treated stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the impact of ipilimumab with vs without gp100 peptides emulsified with Montanide ISA-51 on clinical response in patients with previously treated, HLA-A*0201 positive stage IV melanoma.

Secondary

* Compare the safety/toxicity profile of these regimens in these patients.
* Determine the immunologic response, as measured by in vitro assays using peripheral blood samples, in patients treated with these regimens.
* Determine the response rate after a re-induction regimen for patients who have relapsed after initial response.
* Determine overall survival.

OUTLINE: This is a randomized, open-label study. Patients are stratified according to ECOG performance status (0 vs 1 or 2) and metastases (M1a vs M1 b or M1c). Patients are randomized to 1 of 2 treatment arms.

* Induction phase:

  * Arm I: Patients receive ipilimumab IV over 90 minutes on day 1.
  * Arm II: Patients receive ipilimumab as in arm I. Patients also receive gp100 peptides emulsified in Montanide ISA-51 subcutaneously (SC) on day 1.

In both arms, treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or better for 12 weeks after 4 courses proceed to maintenance phase.

* Maintenance phase:

  * Arm I: Patients receive ipilimumab IV over 90 minutes on day 1.
  * Arm II: Patients receive ipilimumab IV as in arm I and gp100 peptides emulsified in Montanide ISA-51 SC on day 1.

Treatment in both arms begins in approximately week 21 and repeats every 3 months for 8 courses in the absence of disease progression or unacceptable toxicity. Patients who relapse or progress while on maintenance phase undergo re-induction comprising 4 courses of treatment with ipilimumab with or without gp100 peptides emulsified in Montanide ISA-51 as in induction phase. Patients achieving responding disease (complete response, partial response, or stable disease) for 12 weeks after re-induction proceed to the maintenance phase as above for up to 8 courses of treatment.

After completion of study treatment, patients are evaluated for 3 weeks after the last treatment, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 94 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV melanoma

  * HLA-A*0201 positive disease
* Previously treated metastatic disease
* Clinically evaluable and measurable disease
* No mucosal or ocular melanoma
* No evidence of active brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* WBC ≥ 2,500/mm³
* Absolute neutrophil count ≥ 1,000/mm³
* Absolute lymphocyte count ≥ 500/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin ≥ 9 g/dL
* Creatinine < 2.5 mg/dL
* AST ≤ 2 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Bilirubin normal (< 3.0 mg/dL if Gilbert's syndrome is present)
* Hepatitis B surface antigen negative
* HIV negativity
* No hepatitis C virus antibodies
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior malignancy except for any of the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * Superficial bladder cancer
  * Carcinoma in situ of the cervix
  * Any other cancer from which patient has been disease free for > 5 years
* No active immune-mediated disease requiring active therapy with any form of steroid or immunosuppressive therapy
* No documented history of any of the following:

  * Inflammatory bowel disease
  * Regional enteritis
  * Connective tissue disorders, such as systemic lupus erythematosus
  * Rheumatoid arthritis
  * Immune-mediated inflammatory eye disease
  * Sjögren's syndrome
  * Inflammatory neurologic disorder, such as multiple sclerosis
  * Any immune-mediated disease that can cause life-threatening symptoms or severe organ/tissue damage, in the opinion of the principal investigator

    * History of vitiligo or immune-mediated thyroiditis allowed
    * Skin rashes associated with previous therapy allowed provided patient has recovered from treatment-related toxicity to < grade 1
* No active infection
* No systemic hypersensitivity to any of the study drugs

  * History of local reactions (e.g., delayed hypersensitivity or glaucomatous reactions) to Montanide ISA-51 allowed
* No underlying medical condition that, in the opinion of the investigator, would preclude study treatment

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior systemic treatment (6 weeks for nitrosoureas) and recovered
* No prior ipilimumab or gp100 vaccines
* More than 4 weeks since prior steroids
* No concurrent systemic or topical corticosteroids or immunosuppressive agents (e.g., cyclosporine or chemotherapy agents), including steroid enemas, inhaled steroids, or steroid eye drops

  * Hormone-replacement therapy allowed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05

PRIMARY OUTCOMES:
Clinical response

SECONDARY OUTCOMES:
Safety and toxicity
Immunologic response
Response rate
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Principal Investigator — NCI - Surgery Branch

REFERENCES:
- [Background] Downey SG, Klapper JA, Smith FO, Yang JC, Sherry RM, Royal RE, Kammula US, Hughes MS, Allen TE, Levy CL, Yellin M, Nichol G, White DE, Steinberg SM, Rosenberg SA. Prognostic factors related to clinical response in patients with metastatic melanoma treated by CTL-associated antigen-4 blockade. Clin Cancer Res. 2007 Nov 15;13(22 Pt 1):6681-8. doi: 10.1158/1078-0432.CCR-07-0187. Epub 2007 Nov 2. PMID 17982122